CLINICAL TRIAL: NCT06484270
Title: The Effect of Simulation Based Safety Mobilization Program Toward Nurses on Patient Outcomes
Brief Title: Effect of Simulation Based Safety Mobilization Program on Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, pınar dogan, Asst.Prof., Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13579
Record Dates: First submitted 2024-06-12; First posted 2024-07-03 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Patient Outcomes; Simulation Based Learning
Keywords: simulation based learning; patient outcomes; safety mobilization

STUDY DESIGN:
Intervention Model Description: An experimental and follow-up study a pre-test, post-test with control group.
Who Masked: Participant, Care Provider
Masking Description: Participant: patients undergoing surgery in post-op 0 and 1 Care provider: surgical nurses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Nurses receiving simulation-based training Patients receiving care from these nurses
  Interventions: Other: Simulation based safety mobilization program
- Control group (No Intervention): Nurses receiving theoritical education Patients receiving care from these nurses

INTERVENTIONS:
Other: Simulation based safety mobilization program — Nurse participants experienced safe patient mobilization with a simulation-based learning method with a standardized patient for 4 weeks.
  Patient participants were mobilized safely under the supervision of a nurse and the care results were measured.
  Arms: Experimental group

SUMMARY:
The aim of the study was to evaluate the effect of safe mobilization training given to nurses through simulation-based learning method on patient care results.. The main questions it aims to answer are:

Is the safe mobilization training given to nurses by simulation-based learning method effective on the performance of nurses? Is the safe mobilization training given to nurses through simulation-based learning effective on patient outcomes?

Researchers will compare drug ABC to a placebo (a look-alike substance that contains no drug) to see if drug ABC works to treat severe asthma.

Nurse Participants will:

Experimental group: Take simulation based safety mobilization program for 4 weeks Control group: Theoretical education for 1 week (two hours)

Patient Participans will:

He/she mobilized by experimental/control groups nurse and care outcomes are measured for 1 week (once before and after practice)

ELIGIBILITY:
Nurses Inclusion Criteria:

* Agreeing to participate in the study,
* Having no simulation-based learning experience before the study,
* Being a bachelor's degree,
* Being actively working in the data collection process.
* Working in the Surgery Clinic for at least 3 months.

Patient Inclusion Criteria:

* Agreeing to participate in the study,
* Not having a mental or cognitive disease
* Having undergone major surgery

Nurses Exclusion Criteria:

* Be a simulation-based learning experience
* Have less than 3 months of professional experience

Patient Exclusion Criteria:

* Having undergone minor surgery
* Having a mental or cognitive disease

Ages: 22 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Practice performance | one week during the simulation experience
  The performance of nurses in the intervention and control groups during the mobilization experiences was measured with a checklist.
Patient outcomes- Blood pressure | Before and after the patient's first mobilization during a day
  It is measured to determine the effect of mobilization performed by nurses in the intervention and control groups on vital sign-blood pressure.
Patient outcomes-Amount of Wound Drenage (ml) | Before and after the patient's first mobilization during a day
  It is measured to determine the effect of mobilization performed by nurses in the intervention and control groups on surgical field drenage.
Patient outcomes-Satisfaction questionnaire | Before and after the patient's first mobilization during a day
  It is measured to determine the effect of mobilization performed by nurses in the intervention and control groups on satisfaction. This questionaire was evaluated by the patient between 1 and 10 points. 1 being the lowest and 10 being the highest.
Patient outcomes-Pain scale | Before and after the patient's first mobilization during a day
  It is measured to determine the effect of mobilization performed by nurses in the intervention and control groups on pain. This measurement was made with a visual analog scale.This scale was evaluated by the patient between 1 and 10 points. 1 being the lowest and 10 being the highest.
Patient outcomes- Heart rate | Before and after the patient's first mobilization during a day
  It is measured to determine the effect of mobilization performed by nurses in the intervention and control groups on vital signs-heart rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No